CLINICAL TRIAL: NCT00999427
Title: Antiseptic Preparation of the Rectum Prior to Transrectal Prostate Biopsy
Brief Title: Prostate Biopsy Antisepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H09-00289
Record Dates: First submitted 2009-10-15; First posted 2009-10-21 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Infective Complications Post-transrectal Prostate Biopsy
Keywords: Povidone-iodine; prostate cancer; biopsy; transrectal ultrasound; urinary tract infection; fever; sepsis; antisepsis; prevention; complications
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Tract Infections; Fever; Sepsis | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): The randomly selected group of subjects who will receive the intervention. The radiologist performing the transrectal prostate biopsy on these subjects will have a gauze soaked with Povidone-iodine over his/her index finger, and will insert this into the rectum. This gauze will be wiped back and forth across the prostate with the finger at least five times from one lateral margin to the other. This will be allowed to dry for 2 minutes before proceeding with the biopsy.
  Interventions: Drug: Povidone-iodine
- B (No Intervention): The randomly selected group of subjects who will receive the standard of care biopsy without any added intervention.

INTERVENTIONS:
Drug: Povidone-iodine — Povidone-iodine 10% solution. A piece of 10x10 cm gauze soaked in Povidone-iodine 10% solution wrapped around the index finger of the examiner is inserted into the rectum of the subject in arm A. This gauze will be wiped back and forth across the prostate with the finger at least five times from one lateral margin of the prostate gland to the other. The examiner will allow at least 2 minutes to elapse between antisepsis and the insertion of the first needle into the prostate in order to allow the Povidone-iodine to dry.
  Other Names: Betadine solution
  Arms: A

SUMMARY:
During a prostate biopsy, a needle is guided through the rectum into the prostate. Although patients are given antibiotics before the biopsy, there is still a risk of bacteria getting from the rectum into the bladder, prostate and bloodstream during the biopsy. For most surgical procedures, the surgical field is cleaned with antiseptic solution, but this is not common practice for prostate biopsies. In this study patients undergoing prostate biopsy will be randomly assigned to either receive an antiseptic preparation of the rectum or no preparation prior to biopsy, and the rate of infection after the biopsy will be determined.

DETAILED DESCRIPTION:
1. Purpose This research aims to determine the efficacy and safety of cleaning the rectal mucosa with antiseptic solution (Povidone-iodine) prior to transrectal prostate biopsy.
2. Hypothesis We hypothesize that prophylactic cleaning of the rectal mucosa with antiseptic solution prior to transrectal prostate biopsy will decrease the rate of infectious complications after biopsy. We believe that this can be achieved without any significant complications related to the antiseptic solution.
3. Justification Prostate cancer is the most common cancer in men. Since the diagnosis of prostate cancer requires a transrectal prostate biopsy, this procedure is performed frequently. More than 6000 biopsies are performed in British Columbia each year, and more than 1000 are performed at Vancouver General and UBC Hospitals (combined numbers). In these hospitals, the biopsy is performed by the radiologists using transrectal guidance. Subjects receive antibiotic prophylaxis in the form of ciprofloxacin for three days starting one day before the biopsy. They also instill an enema into the rectum a few hours before the biopsy to empty the rectum. Local anesthetic is injected through the rectal mucosa into the periprostatic space prior to the biopsy. Depending on the size of the prostate, between 8 and 12 cores of tissue are remove from the prostate by repetitive passes of the 18 gauge biopsy needle through the anterior rectal wall. Cleaning the rectum with an antiseptic solution prior to biopsy is not routinely practiced and is not considered a current standard of care.

   Despite routine antibiotic prophylaxis, prostate biopsies are associated with a considerable rate of infectious complications. Sepsis after biopsy is described in the literature with an incidence 0.1 to 2.0 %.

   Rate of sepsis has been determined in a retrospective but contemporary study of approximately 4500 biopsies at VGH/UBC to occur with a rate of 0.55% (Lange et al., submitted to Journal of Urology). Less severe but more common adverse events include urinary tract infection and fever, which both occur in approximately 10% of men undergoing biopsy.

   Cleaning the rectum prior to biopsy offers a potential method to decrease the risk of these infectious complications, and we propose the use of Povidone-iodine for this purpose. Surgical site disinfection is standard in most surgical procedures, and Povidone-iodine is a safe antiseptic utilized routinely for the surgical preparation of the body surface as well as mucosal surfaces, including the vagina, mouth and bowel. Park et al. reported that the mean number of colony-forming units decreased 99.9% after Povidone-iodine cleansing of the rectum. Hay et al. reported similar results with Povidone-Iodine enema administration when combined with metronidazole. Povidone-iodine has been shown to significantly reduce bacterial concentrations in the mucosa of the colon and rectum. Brown et al. reported that a Povidone-iodine enema provided a safe and effective means for preventing bacteremia and bacteruria after transrectal prostate biopsy. Furthermore, severe allergic reaction to Povidone-iodine is rare.
4. Objectives

The objectives of this study are:

1. To determine whether cleaning the lining of the rectum with an antiseptic solution before prostate biopsy is effective in decreasing the rate of three outcome variables:

   * Urinary Tract Infection
   * Fever
   * Sepsis
2. To determine at what rate bacteria are found in the rectum prior to biopsy that are resistant to ciprofloxacin.
3. To determine at what rate bacteria are found in the urine after biopsy, with or without rectal cleaning.
4. To determine any adverse reactions to antiseptic solution in the rectum.
5. Research Method All subjects undergoing transrectal prostate biopsy as clinically indicated and determined by the treating Urologist at Vancouver General Hospital and University of British Columbia Hospital will be considered for entry into this trial. If the subject consents to participation, he will be randomized to undergo prostate biopsy with rectal cleaning with antiseptic solution ("treatment" group) or without rectal cleaning ("control" group). A urine sample will be collected before and after biopsy and sent for routine culturing. A rectal swab will be taken before the biopsy (and before rectal cleaning in treatment group) and will be cultured in ciprofloxacin-enriched medium.

   In the treatment group, the radiologist performing the biopsy will wipe the rectal lining overlying the prostate with gauze soaked with Povidone-iodine. Otherwise the biopsy is performed in standard fashion in both groups. After the procedure, the subjects are instructed to measure and record their temperature every 6 hours for 48 hours. A telephone interview is conducted seven days after biopsy to ascertain any adverse events from the biopsy, including whether a temperature ≥38.0˚C was measured.
6. Statistical Analysis The primary outcome in this study will be the rate of urinary tract infection and the rate of fever after biopsy (see definitions below). The rate of sepsis will be measured, but the study will not be powered to detect a difference in the rate of sepsis.

   The rate of UTI and fever is estimated from the literature data at 10% each. A relative reduction of 50% (absolute reduction from 10% to 5%)would be considered clinically significant. With type I & II errors set at 0.05 and 0.2, respectively, and a two-sided test of significance, the necessary sample size is estimated at 435 in each group. Assuming 20% inability to enroll and loss to follow up, the total sample size is 1044.

   Descriptive statistics of baseline parameters will be provided in each group. The mean, median, standard deviation or range of the variables will be computed as applicable. The association between exposure and the defined outcomes will be assessed in univariate analysis. The proportion of each outcome in each group will be compared using the chi square test. Multivariate analysis using logistic regression will be performed to assess effect of variables such as age, number of biopsy cores, individual performing the biopsy and other co-morbidities. A test of interaction will be performed.
7. Definition of Endpoints

   * Urinary tract infection: > 100 million colony forming units per liter in the urine culture obtained48 hours after biopsy.
   * Fever: oral temperature ≥38.0˚C within 48 hours after biopsy.
   * Sepsis(19),(20): positive urine or blood culture plus two or more of the following within 1week of biopsy:

     1. temperature ≥38.0˚C or < 36.0˚C,
     2. heart rate >90 beats/minute,
     3. respiratory rate > 20 breaths/min,
     4. WBC count >12.0 or <4.0 x 10 9/L, or > 0.10 immature forms (bands).
8. Summary of Procedures:

Eligible subjects will be counseled in the office regarding the prostate biopsy as per each physician's routine. This includes instructions for ciprofloxacin prophylaxis (1000 mg of extended release ciprofloxacin daily for three days starting the day before the biopsy) and the use of a fleet enema at home approximately 2 hours before biopsy. The Urologist will also discuss this study with the subject at the same time as he/she orders the biopsy. He/she will ensure that the subject meets the eligibility criteria using a pre-biopsy questionnaire. The subject will be able to take the consent home for further consideration and discussion. It must be signed before the biopsy for the subject to participate in the study.

Each subject will be assigned a study code. At the time of biopsy, subjects will be randomized 1:1 by computer generated random numbers into two groups. The first group ("controls") will undergo biopsy according to the current standard of care, which does not include antiseptic cleaning. The second group ("treatment") will undergo biopsy in the same fashion, but after cleaning the rectal lining with 10% Povidone-iodine.

Before the biopsy is started, the subject is asked to give a midstream urine sample for routine culture. A culture swab is also inserted into the rectum and then cultured in ciprofloxacin-enriched media in order to isolate ciprofloxacin-resistant rectal flora prior to the biopsy.

The control group will undergo the routine biopsy while in the treatment group, the radiologist performing the biopsy will have a gauze soaked with Povidone-iodine over his/her index finger, and will insert this into the rectum. Before this, the Radiologist asks the subject again if he has allergy to Povidone-iodine, shellfish or IVP dye. The gauze will be wiped back and forth across the prostate with the finger at least five times from one lateral margin to the other. The radiologist will allow at least 2 minutes to pass between prep and the insertion of the first needle into the prostate in order to allow the Povidone-iodine to dry. The radiologist will ask the subject to inform the Radiologist if the subject does experience any symptoms of allergic reaction (rash; hives; itching; difficulty breathing; tightness in the chest; swelling of the mouth, face, lips, or tongue ). The 2 minutes will be spent measuring the prostate size using the rectal ultrasound probe. After those two minutes the routine biopsy is done. A second rectal swab for culture will not be taken, as this will likely be negative due to the Povidone-iodine contamination of the swab, and due to the added cost.

All subjects will be discharged from the recovery according to standard care. During the recovery period, a watchful eye is kept on the subjects in the treatment group for developing severe allergic reaction. A crash-cart will be available all the time during the procedure and in the recovery room. Should the subject develop an allergic reaction, the radiologist will take the necessary measures as per the Radiology Department standard of care protocol. The subjects will be asked to provide another midstream urine sample for routine culturing 2 days after the biopsy. This will be grown in conventional media. Subjects will be asked to measure and record their oral temperature once they wake up and just before going to sleep and every 6 hours in between, for 2 days after the procedure. A telephone interview using a post-biopsy questionnaire will be performed with the subject seven days after the biopsy to ascertain any side effects from the biopsy, including whether a temperature ≥38.0˚C was measured.

ELIGIBILITY:
Inclusion Criteria:

* All subjects scheduled at Vancouver General & UBC Hospitals for a transrectal ultrasound guided prostate biopsy are eligible for this study. The indication for biopsy is made according to standard clinical reasoning and judgment, and is not affected by this study.
* All subjects must be willing and able to sign an informed consent and to take the ciprofloxacin prophylaxis before biopsy.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 865 (Actual)
Dates: Start 2009-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Positive urine culture: bacterial growth >100 million colony forming units per litre from mid-stream voided urine sample | 48 hours after biopsy
Fever: oral temperature ≥38.0˚C | within 48 hours of biopsy
Sepsis: patient found to have positive urine culture and/or blood culture plus 2 or more of the following: i. temperature ≥38.0˚C or <36.0˚C ii. heart rate >90 beats/min. iii. respiratory rate >20 breaths/min iv. WBC count >12.0 or <4.0x109/L | within 1 week of biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Peter Black, MD, FRCSC, Principal Investigator — University of British Columbia; S. Larry Goldenberg, MD, FRCSC, Study Director — University of British Columbia; Lindsay Machan, MD, FRCPC, Study Director — University of British Columbia; Martin E. Gleave, MD, FRCSC, Study Chair — University of British Columbia; William Bowie, MD, FRCPC, Study Chair — University of British Columbia; Alan I. So, MD, FRCSC, Study Director — University of British Columbia; Diane Roscoe, MD, FRCPC, Study Director — University of British Columbia; Martin McLoughlin, MD, FRCSC, Study Chair — University of British Columbia; Kourosh Afshar, MD, FRCSC, Study Chair — University of British Columbia; Allen Rowley, MD, FRCPC, Study Chair — University of British Columbia; Alison Harris, MD, FRCPC, Study Chair — University of British Columbia; Anne Buckley, MD, FRCPC, Study Chair — University of British Columbia; Stephen Ho, MD, FRCPC, Study Chair — University of British Columbia; Audrey Spielmann, MD, FRCPC, Study Chair — University of British Columbia; Silvia Chang, MD, FRCPC, Study Chair — University of British Columbia; Zeid AbuGhosh, MD, FEBU, Study Chair — University of British Columbia
Locations (3):
- Canada (3):
  - Department of Urologic Sciences, Gordon & Leslie Diamond Health Care Centre, Vancouver, British Columbia
  - Radiology Department - UBC Hospital, Vancouver, British Columbia
  - Radiology Department - Vancouver General Hospital, Vancouver, British Columbia